CLINICAL TRIAL: NCT05682157
Title: Use of the Paula Method of Muscle Exercises Among Patients With Low Anterior Resection Syndrome After Sphincter-sparing Rectal Resection Using an Integrative Approach
Brief Title: Paula Method of Exercises in Patients With LARS Syndrome:Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCT-PAULA-LARS-HMO-CTIL
Record Dates: First submitted 2022-12-27; First posted 2023-01-12 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Low Anterior Resection Syndrome
Keywords: Paula Method; Sphincter sparing rectal resection; Anal incontinence; Rectal Cancer
MeSH Terms: conditions — Low Anterior Resection Syndrome; Encopresis; Rectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Paula Method (Experimental): 12 weeks of the Paula Method of muscle exercises with standard care
  Interventions: Other: Paula Method of muscle exercises
- Standard Care (No Intervention): standard care

INTERVENTIONS:
Other: Paula Method of muscle exercises — 12 weekly sessions of Paula Method of exercise
  Arms: Paula Method

SUMMARY:
Sphincter sparing rectal resection surgery, either total mesorectal excision (TME) with a temporary loop ileostomy or partial mesorectal excision (PME), is the mainstay of rectal cancer treatment , however, these treatments are associated with the development of Low anterior resection syndrome (LARS). This syndrome is characterized by a constellation of symptoms such as fecal frequency, urgency and clustering of bowel movements and can lead to fecal and flatus incontinence. There is no gold standard therapy designed to treat the root cause of the problems associated with LARS. Paula Method of exercises, based on the theory that the body has the natural ability to self-heal and that all sphincter muscles in the body affect one another other and thus, exercising one healthy region can positively impact another. The purpose of this study is to evaluate the usefulness of the Paula Method of exercises in patients post sphincter sparing rectal resection surgery with LARS Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* patients 6-18 months post restorative surgery (either resection with a primary functional anastomosis or after the closure of a temporary ileostomy following curative surgery for rectal cancer) and, if applicable, at least one month post last adjuvant chemotherapy treatment
* LARS score of 21 or greater
* age 18 or older
* able to read and write in Hebrew or English
* able and willing to comply with the study requirements.

Exclusion Criteria:

* Chronic anal incontinence prior to surgery
* inability to perform exercises due to cognitive or physical limitations
* actively engaged in pelvic floor muscle exercises
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in LARS score | 12 weeks
  Comparison of the change in LARS score from baseline to the completion of 12 weeks of the intervention (within and between groups).

CONTACTS AND LOCATIONS:
Overall Officials: Noam Shussman, MD, Principal Investigator — Hadassah Medical Organization
Locations (2):
- Israel (2):
  - Hadassah Medical Organization, Jerusalem
  - Rabin Medical Center, Petah Tikva

IPD SHARING:
Plan to Share IPD: No